CLINICAL TRIAL: NCT04910984
Title: Developing an Artificial Intelligence Chatbot to Promote HIV Testing
Brief Title: Developing a Chatbot to Promote HIV Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: University of Malaya (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2000027864; 1R21AI152927-01A1 (NIH)
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: HIV testing; PrEp; HIV care; Chatbot; MSM
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chatbot group (Experimental)
  Interventions: Behavioral: Chatbot messages
- TAU group (Placebo Comparator)
  Interventions: Behavioral: Attention-matched educational materials

INTERVENTIONS:
Behavioral: Chatbot messages — Automated personalized messages containing HIV testing-related information, motivation and skills
  Arms: Chatbot group
Behavioral: Attention-matched educational materials — Attention-matched educational materials manually sent by our research assistant. These educational materials will be retrieved from CDC and WHO websites and curated into short articles (<200 words) and pictures. All educational materials will be screened by HIV experts from University of Malaya to ensure accuracy before being sent to participants.
  Arms: TAU group

SUMMARY:
In this study, the feasibility of a Chatbot in promoting HIV testing in a pilot RCT with 80 men who have sex with men in Kuala Lumpur, Malaysia will be studied. Participants will be randomized to Chatbot or treatment as usual (TAU) groups. Participants in the intervention group will receive automated personalized messages containing HIV testing-related information, motivation and skills.

DETAILED DESCRIPTION:
After informed consent, participants will be randomly assigned to Chatbot or TAU groups using stratified randomization by age. Participants in TAU will receive attention-matched educational materials manually sent by the research assistant. Participants in the intervention group will receive an automated personalized question message (root-node message) from the Chabot. In each round of the interactive communication, the Chatbot will provide automated personalized messages containing HIV testing-related information, motivation and skills based on participants' answers and will continuously update over time. Participants will be observed over 180 days with responses and interactions stored on a HIPAA-compliant and protected cloud. An independent assessment of recent testing and reasons why will be sent by link to both TAU and intervention groups using a link to a Qualtrics survey housed on REDCap at baseline and after 90 and 180 days. After 180 days, the RA will send an additional REDCap survey to intervention participants to assess the feasibility of the Chabot to measure 4 key elements: acceptability, practicality, demand, and adaptation.

ELIGIBILITY:
Inclusion Criteria:

* cis-gender male
* 18+ years;
* had condomless sex with men in the past 6 months
* has a smartphone
* speaks Bahasa Malay or English.

Exclusion Criteria:

* Not able to read Malay or English

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-07-20 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in HIV testing | 30 days, 60 days, 90 days, 120 days, 150 days, and 180 days
  The efficacy of the Chatbot versus TAU with HIV testing as the primary outcome will be measured. The primacy efficacy outcome is the proportion of MSM who get tested within 180 days. This will be measured every 30 days by asking if MSM tested for HIV in the past 30 days.

SECONDARY OUTCOMES:
Recruitment rate | 180 days
  The number of participants contacted divided by the number of participants who signed the consent form
Completion rate | 180 days
  The number of participants who signed the consent form divided by the number of participants who completed the study
Interaction time | 180 days
  The time of the interaction between participants and Chatbot
Interaction frequency | 180 days
  The frequency of the interaction between participants and Chatbot

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A. Wickersham, PhD, Principal Investigator — Yale University
Locations (1):
- University of Malaya, Kuala Lumpur, Jalan Pantai Baharu, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided